CLINICAL TRIAL: NCT03006913
Title: Comparison of 3 Modes of Genetic Counseling in High-Risk Public Hospital
Brief Title: Comparison of 3 Modes of Genetic Counseling in High-Risk Public Hospital Patients
Acronym: GC3Modes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of California, Davis (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCSF-GC3-2021; R01CA197784-01A1 (NIH)
Record Dates: First submitted 2016-11-16; First posted 2016-12-30 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Genetic Counseling
Keywords: Genetic counseling modes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Randomization to counseling: In-person (Active Comparator): Behavioral: Comparing genetic counseling modes.
  Interventions: Behavioral: In-person
- Randomization to counseling: By phone (Active Comparator): Behavioral: Comparing genetic counseling modes.
  Interventions: Behavioral: By phone
- Randomization to counseling: By video (Active Comparator): Behavioral: Comparing genetic counseling modes.
  Interventions: Behavioral: By video

INTERVENTIONS:
Behavioral: In-person — At all sites, patients randomized to/preferring in-person counseling will meet with a counselor.
  Arms: Randomization to counseling: In-person
Behavioral: By phone — Patients in the phone arm will receive a scheduled call at their home.
  Arms: Randomization to counseling: By phone
Behavioral: By video — Because low income patients are not likely to have video conference capability at home, this service will be offered at all three hospitals, and patients will have scheduled appointments to come to the hospital to receive counseling delivered through a computer.
  Arms: Randomization to counseling: By video

SUMMARY:
Using mixed methods, investigators will conduct a multicenter partially randomized preference noninferiority trial with high-risk English-, Spanish-, and Cantonese-speaking patients assigned by (1) patients´ preference or (2) randomization to three counseling modes: (a) in-person; (b) phone; or (c) video conference. A total of 600 patients will complete counseling and 540 will complete the final survey. Baseline and post-counseling surveys will use validated measures (adapted for literacy and language) of study outcomes. All counseling sessions will be audio-taped. A sample of 90 tapes will be analyzed for counseling content and to identify 30 participants for in-depth interviews and analysis triangulating all forms of data. Genetic counselors will be interviewed in depth to elicit their perceptions of the strengths and limitations of each counseling mode.

DETAILED DESCRIPTION:
Specific Aims.

The specific aims of this mixed methods study are:

Aim 1. Compare the effectiveness of 3 modes of genetic counseling in a diverse sample of patients at high risk for HBOC in 3 public hospitals. Conduct a multicenter partially randomized preference noninferiority trial with high-risk patients assigned by (a) randomization to three counseling modes: in-person, phone, video conference; or (b) patients´ preference. Utilize validated measures of study outcomes adapted as needed for literacy and language. Recognizing that some potential participants may have a strong preference for one counseling mode, after explaining the study design and obtaining informed consent, participants will be asked if they have such a preference. Those who do will be offered that mode, and those who do not will be randomized. Randomization will be stratified according to hospital and personal history of breast cancer in order to ensure that there is no imbalance in important factors that may be associated with outcome.

Aim 2. Explore inductively and qualitatively variation in patients' genetic counseling experiences and understandings, genetic counselor satisfaction and perceptions, counseling session similarities and differences, and implications of organizational context across three modes of genetic counseling.

Aim 3 employs inductive, qualitative methods to explore in depth the cases of 30 patients using their pre- and post-counseling survey responses, audio tapes of their counseling session, and in-depth interviews to explore questions common to all respondents and those specific to what was learned about the individual from the other data sources. In-depth interviews will also be conducted with genetic counselors.

Study Design:

Using mixed methods, investigators will conduct a multicenter partially randomized preference noninferiority trial with high-risk English-, Spanish-, and Cantonese-speaking patients assigned by (1) patients´ preference or (2) randomization to three counseling modes: (a) in-person; (b) phone; or (c) video conference. A total of 600 patients will complete counseling and 540 will complete the final survey. Baseline and post-counseling surveys will use validated measures (adapted for literacy and language) of study outcomes. All counseling sessions will be audio-taped. A sample of 90 tapes will be analyzed for counseling content and to identify 30 participants for in-depth interviews and analysis triangulating all forms of data. Genetic counselors will be interviewed in depth to elicit their perceptions of the strengths and limitations of each counseling mode.

Investigators' mixed methods combine a multicenter partially randomized preference noninferiority trial with inductive methods that embed this research in the real world of public health system patients. This is practice-based research, designed to emphasize external validity, (relevance and generalizability that enhance translation into actual use), as well as internal validity. The purpose of a non-inferiority trial is to compare an intervention to an active control or standard treatment when the intervention is not expected to have superior efficacy, but to have other benefits, e.g., greater convenience or fewer side effects. In the case of genetic counseling, in- person counseling is the standard of care, with well-documented efficacy.4 Since video and telephone counseling do not offer a more personalized approach or more pertinent content than in-person counseling, it seems unlikely that either mode would produce superior psychosocial outcomes or greater knowledge gains; similarly, investigators do not expect telephone counseling to be more efficacious than video counseling.

The gold standard for assessing the effectiveness of interventions is the randomized clinical trial; yet patients who have a strong preference for one of the intervention conditions may decline to participate, which is a threat to external validity, or (if randomized) participate half-heartedly or drop out, threatening internal validity. Investigators will address this issue with a partially randomized preference trial in which patients with a strong preference are assigned to their preferred treatment (i.e., intervention condition) and those without a strong preference are randomized. This study design enables comparison of treatment outcomes among patients who receive their preferred treatment (the desired real world situation) and ascertainment of the effects of preference-as well as the evaluation of treatment outcomes in a randomized trial. However, comparisons involving preference participants are subject to confounding, since patients who prefer a particular treatment may differ in ways that affect outcome. In analyses involving preference participants it is possible to reduce confounding substantially using covariate adjustment. Nevertheless, because residual confounding may be present, preference participant outcomes should be considered observational data.

Investigators will blend qualitative and quantitative, deductive and inductive methods using varied forms of data from in-depth interviews, surveys, and audio taped observations. This will allow us to address our central question from different perspectives triangulated in the analysis for a rich understanding of patient-counselor- institution relationships most of which are too complex to describe using one dimension alone (e.g., cognitive understanding captured in surveys). While the randomized trial is the gold standard for comparative effectiveness, it cannot answer questions such as what it is about the counseling interaction that was reassuring or anxiety-provoking to a patient? what techniques enabled a patient to recall important points? or what about the conversation precluded such recall? It is only by embedding the survey data in open-ended inductive exploration and audio observations that investigators can determine if a counselor provided too much information to a low-literacy patient, or alternatively used plain language to emphasize key points, checking frequently for patient comprehension. Importantly, was the counselor able to do this as well by phone or video? Thus, mixed methods illuminates important dynamics that informants may not be consciously aware of.

ELIGIBILITY:
Inclusion Criteria:Eligible participants include patients who

* visit the mammography, high risk or oncology clinics at Contra Costa County, Highland or SFGH hospitals,
* are referred to genetic counseling services at SFGH by a community clinic through the E-Referral system or are considered to be high risk based on their breast/ovarian cancer genetics Referral Screening Tool (RST) score (≥ 2 checks)
* speak English, Spanish, or Cantonese

Investigators will also include two genetic counselors who provide services at SFGH and UCSF.

Exclusion Criteria:

* do not speak English, Spanish, or Cantonese;
* are age 17 and under; and
* don't have a family history of cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1273 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Differences in change scores among three counseling modes: Breast Cancer Knowledge Scale | One week post counseling
  Will measure knowledge of hereditary breast cancer information before and after delivery of counseling modes.
Differences in change scores among three counseling modes: Impact of Events Scale | One week post counseling
  Will measure cancer-specific distress before and after delivery of counseling modes.

SECONDARY OUTCOMES:
Differences in change scores among three counseling modes: Decisional Conflict Scale | One week post counseling
  Will measure decisional conflict before and after implementation of counseling modes.
Differences in change scores among three counseling modes: Perceived Stress Scale | One week post counseling
  Will measure general perceptions of stress before and after implementation of counseling modes.
Differences in change scores among three counseling modes: Breast/Ovarian Cancer Risk Perception and Worry Scale | One week post counseling
  Will measure breast cancer and ovarian cancer risk perception and worry before and after implementation of counseling modes.
Differences in change scores among three counseling modes: Perceptions of Risks and Benefits of Genetic Counseling Scale | One week post counseling
  Will measure perceptions of risks and benefits of genetic counseling before and after implementation of counseling modes.
Differences in change scores among three counseling modes: Genetic Counseling Satisfaction Scale | One week post counseling
  Will measure genetic counseling satisfaction before and after implementation of counseling modes.

CONTACTS AND LOCATIONS:
Overall Officials: Rena J. Pasick, DrPH, Principal Investigator — University of California, San Francisco; Galen Joseph, PhD, Principal Investigator — Universidad de California, San Francisco; Claudia S Guerra, MSW, Study Director — University of California, San Francisco
Locations (3):
- United States (3):
  - Contra Costa Regional Medical Center Health Services, Martinez, California
  - Highland General Hospital, Oakland, California
  - San Francisco General Hospital, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King MC, Marks JH, Mandell JB; New York Breast Cancer Study Group. Breast and ovarian cancer risks due to inherited mutations in BRCA1 and BRCA2. Science. 2003 Oct 24;302(5645):643-6. doi: 10.1126/science.1088759. PMID 14576434
- [Background] Whittemore AS, Gong G, John EM, McGuire V, Li FP, Ostrow KL, Dicioccio R, Felberg A, West DW. Prevalence of BRCA1 mutation carriers among U.S. non-Hispanic Whites. Cancer Epidemiol Biomarkers Prev. 2004 Dec;13(12):2078-83. PMID 15598764
- [Background] Anglian Breast Cancer Study Group. Prevalence and penetrance of BRCA1 and BRCA2 mutations in a population-based series of breast cancer cases. Anglian Breast Cancer Study Group. Br J Cancer. 2000 Nov;83(10):1301-8. doi: 10.1054/bjoc.2000.1407. PMID 11044354
- [Background] Nelson HD, Pappas M, Zakher B, Mitchell JP, Okinaka-Hu L, Fu R. Risk assessment, genetic counseling, and genetic testing for BRCA-related cancer in women: a systematic review to update the U.S. Preventive Services Task Force recommendation. Ann Intern Med. 2014 Feb 18;160(4):255-66. doi: 10.7326/M13-1684. PMID 24366442
- [Background] Schwartz MD, Valdimarsdottir HB, Peshkin BN, Mandelblatt J, Nusbaum R, Huang AT, Chang Y, Graves K, Isaacs C, Wood M, McKinnon W, Garber J, McCormick S, Kinney AY, Luta G, Kelleher S, Leventhal KG, Vegella P, Tong A, King L. Randomized noninferiority trial of telephone versus in-person genetic counseling for hereditary breast and ovarian cancer. J Clin Oncol. 2014 Mar 1;32(7):618-26. doi: 10.1200/JCO.2013.51.3226. Epub 2014 Jan 21. PMID 24449235
- [Background] Kinney AY, Butler KM, Schwartz MD, Mandelblatt JS, Boucher KM, Pappas LM, Gammon A, Kohlmann W, Edwards SL, Stroup AM, Buys SS, Flores KG, Campo RA. Expanding access to BRCA1/2 genetic counseling with telephone delivery: a cluster randomized trial. J Natl Cancer Inst. 2014 Nov 5;106(12):dju328. doi: 10.1093/jnci/dju328. Print 2014 Dec. PMID 25376862
- [Background] Madlensky L. Is it time to embrace telephone genetic counseling in the oncology setting? J Clin Oncol. 2014 Mar 1;32(7):611-2. doi: 10.1200/JCO.2013.53.8975. Epub 2014 Jan 21. No abstract available. PMID 24449232
- [Background] Hall MJ, Olopade OI. Disparities in genetic testing: thinking outside the BRCA box. J Clin Oncol. 2006 May 10;24(14):2197-203. doi: 10.1200/JCO.2006.05.5889. PMID 16682739
- [Background] Narod SA, Foulkes WD. BRCA1 and BRCA2: 1994 and beyond. Nat Rev Cancer. 2004 Sep;4(9):665-76. doi: 10.1038/nrc1431. PMID 15343273
- [Background] Forman AD, Hall MJ. Influence of race/ethnicity on genetic counseling and testing for hereditary breast and ovarian cancer. Breast J. 2009 Sep-Oct;15 Suppl 1:S56-62. doi: 10.1111/j.1524-4741.2009.00798.x. PMID 19775331
- [Background] Armstrong K, Micco E, Carney A, Stopfer J, Putt M. Racial differences in the use of BRCA1/2 testing among women with a family history of breast or ovarian cancer. JAMA. 2005 Apr 13;293(14):1729-36. doi: 10.1001/jama.293.14.1729. PMID 15827311
- [Background] Sussner KM, Jandorf L, Thompson HS, Valdimarsdottir HB. Interest and beliefs about BRCA genetic counseling among at-risk Latinas in New York City. J Genet Couns. 2010 Jun;19(3):255-68. doi: 10.1007/s10897-010-9282-4. Epub 2010 Feb 12. PMID 20151317
- [Background] Halbert CH, Kessler L, Stopfer JE, Domchek S, Wileyto EP. Low rates of acceptance of BRCA1 and BRCA2 test results among African American women at increased risk for hereditary breast-ovarian cancer. Genet Med. 2006 Sep;8(9):576-82. doi: 10.1097/01.gim.0000237719.37908.54. PMID 16980814
- [Background] Karliner LS, Napoles-Springer A, Kerlikowske K, Haas JS, Gregorich SE, Kaplan CP. Missed opportunities: family history and behavioral risk factors in breast cancer risk assessment among a multiethnic group of women. J Gen Intern Med. 2007 Mar;22(3):308-14. doi: 10.1007/s11606-006-0087-y. PMID 17356960
- [Background] Joseph G, Guerra C. To worry or not to worry: breast cancer genetic counseling communication with low-income Latina immigrants. J Community Genet. 2015 Jan;6(1):63-76. doi: 10.1007/s12687-014-0202-4. Epub 2014 Aug 23. PMID 25148879
- [Background] Green LW, Glasgow RE. Evaluating the relevance, generalization, and applicability of research: issues in external validation and translation methodology. Eval Health Prof. 2006 Mar;29(1):126-53. doi: 10.1177/0163278705284445. PMID 16510882
- [Background] D'Agostino RB Sr, Massaro JM, Sullivan LM. Non-inferiority trials: design concepts and issues - the encounters of academic consultants in statistics. Stat Med. 2003 Jan 30;22(2):169-86. doi: 10.1002/sim.1425. PMID 12520555
- [Background] Vig HS, Wang C. The evolution of personalized cancer genetic counseling in the era of personalized medicine. Fam Cancer. 2012 Sep;11(3):539-44. doi: 10.1007/s10689-012-9524-8. PMID 22419176
- [Background] Lea DH, Kaphingst KA, Bowen D, Lipkus I, Hadley DW. Communicating genetic and genomic information: health literacy and numeracy considerations. Public Health Genomics. 2011;14(4-5):279-89. doi: 10.1159/000294191. Epub 2010 Apr 20. PMID 20407217
- [Background] Cohen SA, Marvin ML, Riley BD, Vig HS, Rousseau JA, Gustafson SL. Identification of genetic counseling service delivery models in practice: a report from the NSGC Service Delivery Model Task Force. J Genet Couns. 2013 Aug;22(4):411-21. doi: 10.1007/s10897-013-9588-0. Epub 2013 Apr 25. PMID 23615968
- [Background] Squiers L, Peinado S, Berkman N, Boudewyns V, McCormack L. The health literacy skills framework. J Health Commun. 2012;17 Suppl 3:30-54. doi: 10.1080/10810730.2012.713442. PMID 23030560